CLINICAL TRIAL: NCT06558175
Title: A Safety and Efficacy Trial of Reirradiation Dose Escalation in Thoracic Cancers: Re-evaluating Previous Dose and Allowing Increasing Recovery (REPAIR)
Brief Title: Reirradiation Dose Escalation in Thoracic Cancers
Acronym: REPAIR
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ReDA 14927
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Thoracic Cancer; Lung Cancer; Esophageal Cancer
Keywords: Re-irradiation; Toxicity; Dose escalation; Oncology
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms; Neoplasms | interventions — Radiosurgery; Radiotherapy

STUDY DESIGN:
Intervention Model Description: This multi-institution phase I dose-escalation study for patients undergoing thoracic re-irradiation will use a time-to-event continual reassessment method (TITE-CRM).
  Accrual will start at level 1 (recovery factor = 10% at 6 months + 0.75% per month thereafter). Patients will be assigned to recovery factors using the TITE-CRM model. The model will use all available information from previously accrued patients to assign the highest dose with a predicted risk of grade 3-5 toxicity of 35% or less.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recovery factor levels (Experimental): Radiation therapy - recovery factor levels Level 1: 6 months (10%) and 0.75%/month Level 2: 6 months (15%) and 0.75%/month Level 3: 6 months (15%) and 1.00%/month Level 4: 6 months (20%) and 1.00%/month Level 5: 6 months (20%) and 1.25%/month Level 6: 6 months (25%) and 1.40%/month
  Interventions: Radiation: stereotactic body radiation therapy (SBRT)

INTERVENTIONS:
Radiation: stereotactic body radiation therapy (SBRT) — Patients will be assigned to treatment doses using the TITE-CRM model.
  Other Names: Radiation therapy

SUMMARY:
This is a study involving patients with recurrence, metastasis, or new primary malignancies in the thorax requiring radiation and who have previously received radiotherapy to the thorax, where re-irradiation is expected to exceed the dose constraints used for de novo treatments.

Currently, when this group of patients needs another set of radiotherapy, there is a dose limitation based on a percentage of the previous treatment's dose. However, this dose often limits the effectiveness of repeated treatment, with little scientific support for such. Therefore, this study aims to determine the maximally tolerated dose of reirradiation in the thorax, with dose escalation implemented by sequentially increasing the normal tissue recovery factors (i.e. repair factors) to the previously delivered dose.

Using a recovery factor equation associated with a 35% or lower rate of grade 3-5 treatment-related toxicity occurring within 1 year of treatment, accrual will start at level 1 (recovery factor = 10% at 6 months + 0.75% per month thereafter). Patients will be assigned to recovery factors using the TITE-CRM model. The model will use all available information from previously accrued patients to assign the highest dose with a predicted risk of grade 3-5 toxicity of 35% or less.

DETAILED DESCRIPTION:
The REPAIR trial aims to identify the magnitude of radiation recovery in the thorax and enable safe reirradiation dose escalation. The trial will provide critical information to support shared-decision making and ensure the risk-benefit trade-offs of reirradiation align with each patient's wishes. In addition, the data from this study will be informative in guiding subsequent studies on the use of reirradiation for other sites (such as the brain, abdomen, and pelvis) and to inform future re-irradiation trials. The objective of this phase I study is to determine the safety of dose escalation via recovery factors applied against previously delivered doses for patients receiving thoracic reirradiation.

This study will use a time-to-event continual reassessment method (TITE-CRM). The study design is based on previous thoracic dose escalation trials.

The primary endpoint of this study is the maximally tolerated dose (MTD) of thoracic reirradiation, implemented by sequentially increasing the normal tissue recovery factors applied to the previously delivered dose. The MTD is the recovery factor equation associated with a ≤ 35% rate of grade 3-5 pre-specified treatment-related toxicity occurring within 1 year of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of malignancy, with disease in the thorax requiring re-irradiation for any treatment intent. This may include primary lung cancer of any type, esophageal cancer, recurrences, and/or metastasis from any primary. The intrathoracic disease at the time of enrollment does not itself require a biopsy if a prior biopsy has been obtained at that location or another body site. If the risk of biopsy is unacceptable and there is no prior confirmation of malignancy even at the time of the initial course of radiation, enrollment is permitted provided that the case is discussed at a multidisciplinary tumor board or peer-review rounds.
* Must have received prior photon thoracic radiotherapy ≥ 6 months ago
* Life expectancy > 6 months.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Age ≥ 18 years
* The current radiation course, when added to the previous radiation doses, exceeds the normal tissue constraints used for de novo treatments for esophagus, heart, lungs, trachea, bronchus, great vessels, or brachial plexus. Forgiveness of the previous dose (i.e. reduction of the previous dose in the cumulative dose calculation) is required to meet constraints. Submission of a pre-plan summary showing the estimated accumulation of current and previously delivered doses is required for registration.

Exclusion Criteria:

* Persistent toxicity from previously delivered radiation therapy
* Prior development of symptomatic radiation pneumonitis or immunotherapy-related pneumonitis from previous treatment, even if resolved
* Cumulative radiation dose for all organs-at-risk is already below dose constraints without a recovery factor applied, or with a recovery factor less than the current dose level of the trial. This will be confirmed by the enrolling team after the planning is completed.
* The reirradiation dose-limiting structure is expected to be spinal cord, chest wall, and/or stomach.
* Any prior thoracic radiotherapy < 6 months ago; OR prior thoracic radiotherapy delivered twice daily (compensation for holiday breaks are OK), thoracic radiotherapy delivered by brachytherapy, radionuclides, proton beams, or electron beams.
* Plans for patient to receive daily adaptive radiotherapy in current plan (computed tomography or magnetic resonance based).
* Plans for the patient to receive other local therapy (including standard fractionated radiotherapy and/or surgery) while on this study, except at disease progression.
* Concurrent systemic therapy (i.e. on the same days as radiation) is not allowed, EXCEPT for patients being treated for intrathoracic lung cancer (NSCLC or SCLC) with curative intent.
* For other patients receiving systemic therapy, they are still eligible for enrollment as long as there is a break in systemic therapy during the course of radiation. For example, if a patient has been on palliative pemetrexed and is planning to continue, they can still be enrolled and would continue to receive pemetrexed; reirradiation would be delivered between cycles, possibly requiring a break in systemic therapy. See Section 6.9 for further details.
* Prior surgical intervention that has significantly changed the position of an organ-at-risk that is expected to be a dose-limiting structure.
* Pregnancy
* The following autoimmune and connective tissue diseases will be excluded: Scleroderma and Systemic lupus erythematosus.
* Patients with interstitial lung disease (ILD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
Maximally tolerated dose (MTD) | occurring within 1 year of treatment
  MTD of radiotherapy for thoracic tumors. The MTD is the dose of radiotherapy associated with a <35% rate of grade 3-5 toxicity occurring within 1 year of treatment.

SECONDARY OUTCOMES:
Time to progression | 1-5 years
  Progression of treated disease
Time to distant metastases | 1-5 years
  Time to distant metastases
Progression-Free Survival | 1-5 years
  Progression-Free Survival
Overall survival | 1-5 years
  Overall survival
Patient reported outcome | Before treatment and at 3, 6, 9, 12, 18, 24, 36, 48, and 60 months
  Functional Assessment of Cancer Therapy: Lung (FACT-L)
Quality of Life - EuroQol 5-dimension 5-level | Before treatment and at 3, 6, 9, 12, 18, 24, 36, 48, and 60 months
  EuroQol 5-dimension 5-level

CONTACTS AND LOCATIONS:
Overall Officials: David Palma, MD,PhD,FRCPC, Principal Investigator — London Health Science Centre

IPD SHARING:
Plan to Share IPD: No